CLINICAL TRIAL: NCT00647166
Title: Evaluation of a New Treatment Strategy for Patients With Microscopic Polyangiitis, Polyarteritis Nodosa or Eosinophilic Granulomatosis With Polyangiitis (Churg Strauss Syndrome) Without Poor Prognosis Factors
Brief Title: Association Corticosteroid/Azathioprine in Microscopic Polyangiitis/ Polyarteritis Nodosa or Eosinophilic Granulomatosis With Polyangiitis (Churg Strauss Syndrome)
Acronym: CHUSPAN2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P 060243
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: MPA; PAN or EGPA With FFS=0; At Diagnosis or Within the First 15 Days Following Initiation of Corticosteroids
Keywords: Vasculitis; Polyarteritis nodosa (PAN); Microscopic polyangiitis (MPA); Eosinophilic granulomatosis with polyangiitis (EGPA); Churg Strauss syndrome (CSS); Azathioprine
MeSH Terms: conditions — Polyarteritis Nodosa; Vasculitis; Microscopic Polyangiitis; Churg-Strauss Syndrome | interventions — Adrenal Cortex Hormones; Azathioprine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Drug: corticosteroid and azathioprine
  Interventions: Drug: corticosteroid and azathioprine
- 2 (Placebo Comparator): Drug: corticosteroid and placebo
  Interventions: Drug: corticosteroid and placebo

INTERVENTIONS:
Drug: corticosteroid and azathioprine — * Corticosteroid 1 mg/kg/day with a conventional decrease dose
  * Azathioprine : 2 mg/kg/day during one year in 2 to 3 times a day by oral route
  Arms: 1
Drug: corticosteroid and placebo — * Corticosteroid 1 mg/kg/day with a conventional decrease dose
  * Placebo : 2 mg/kg/day during one year in 2 to 3 times a day by oral route
  Arms: 2

SUMMARY:
To determine whether a combination of corticosteroids and azathioprine can achieve a higher remission rate and a lower subsequent relapse rate in patients with newly-diagnosed microscopic polyangiitis, polyarteritis nodosa or eosinophilic granulomatosis with polyangiitis (Churg Strauss syndrome) with no poor prognosis factor (FFS=0), and without significantly increasing the rate of adverse events, as compared to corticosteroids alone. The study hypothesis is a reduction of the absolute risk of treatment failure or relapse within the first 24 months following initiation of therapy of least 25%.

DETAILED DESCRIPTION:
Patients with new diagnosis of 1) microscopic polyangiitis, polyarteritis nodosa or eosinophilic granulomatosis with polyangiitis (Churg Strauss syndrome) and 2) without any factor of poor prognosis according to the French five factors score (FFS - including creatininemia >140µmol/l, proteinuria >1 g/24 h, specific gastro-intestinal involvement, specific cardiomyopathy, and CNS involvement) can be included at diagnosis or within the first 15 days following initiation of corticosteroids. Treatment is randomly assigned, centrally, and received in a double-blinded fashion. It consists in a combination of azathioprine (2 mg/kg/day) and corticosteroids (starting at 1 mg/kg/day for 3 weeks then progressively tapered over a mean of 50 weeks, varying according to patient's weight) or, for the control group, the same corticosteroid therapy plus placebo. Duration of azathioprine or placebo is 12 months, and patients are followed for 12 additional months, yielding in a total duration of the protocol of 24 months after entry for each patient. End point is the number of patients who achieve sustained remission and who do not suffer a relapse during the 24 months of the study protocol. Based on the results of the early CHUSPAN trial for similar patients treated with corticosteroids alone, the cumulative rate of failures and relapses can be estimated at 40% at 24 months. The primary hypothesis of the CHUSPAN 2 is a reduction by at least 25% for the rate of this combined parameter of remission-treatment failure and relapse at 24 months. Based on this hypothesis, using a bilateral test, with a significance level of 5%, a beta level of 80% and an estimated 5% of lost-of-follow-up, 104 patients must be included. Secondary end points include the initial remission rate (independently of subsequent relapses), rate of adverse events and their severity according to the WHO toxicity grading system, number of deaths, number of patients who could not be weaned of corticosteroids, area under the curve for corticosteroids, and different scales, such as BVAS (activity of the disease), VDI (damage), HAQ, SF36, ADL and the evaluation of the need for health care facilities.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients
* aged over 18 years
* new diagnosis of microscopic polyangiitis, polyarteritis nodosa or eosinophilic granulomatosis with polyangiitis (Churg Strauss syndrome), satisfying ACR 1990 and/or Chapel Hill Nomenclature criteria (positive biopsy is not mandatory providing those criteria are fulfilled)
* with no factor of poor prognosis according to the French five factors score (FFS=0)
* at diagnosis or within the first 21 days following initiation of corticosteroids
* signed information and consent form
* patients covered by Health Insurance
* having had a baseline physical examination

Exclusion Criteria:

* patients with microscopic polyangiitis, polyarteritis nodosa or eosinophilic granulomatosis with polyangiitis (Churg Strauss syndrome) with one or more factor(s) of poor prognosis according to the French five factors score (FFS ≥ 1)
* patients with polyarteritis nodosa with ANCA, not satisfying the criteria for microscopic polyangiitis
* patients with clinically overt alveolar hemorrhage or respiratory distress syndrome
* patient treated with corticosteroids for more than 15 days or already receiving another immunosuppressant
* relapsing vasculitis
* other vasculitis, especially secondary vasculitides
* vasculitis secondary or associated with a viral infection, such as hepatitis B or C virus, or HIV
* malignancy
* pregnancy and breast feeding,women of child-bearing age not willing or with contra-indication to receive contraception
* contra-indication to any of the study agents
* need to continue allopurinol for those patients taking allopurinol
* consent deny or inability to receive information and give consent
* participation in another concomitant therapeutic trial
* no affiliation to any of the general French health care system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-05; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
combined rate of remission-treatment failures and minor or major relapses at 24 months | 24 months

SECONDARY OUTCOMES:
initial remission rate (independently of subsequent relapse) | 24 months
number of patients who have a minor or major relapse | 24 months
number of serious treatment-related adverse effects | 24 months
number of patients with at least one treatment-related adverse effect | 24 months
severity of treatment-related effects according to the WHO toxicity grading system (grades 1 to 4; grades 3 and 4 for the severity) | 24 months
number of deaths and causes | 24 months
number of patients who could not be weaned of corticosteroids and dose required | 24 months
area under the curve for corticosteroids | 24 months
different scales, such as BVAS (activity of the disease), VDI (damage), HAQ, SF36, ADL and the evaluation of the need for health care facilities. | 24 months
number of flares with or without asthma and/or eosinophilia (only for EGPA analysis) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Loic Guillevin, MD, PhD, Study Director — French Vasculitis Study Group
Locations (1):
- Hopital Cochin Pôle de Médecine UF Médecine Interne, Paris, France

REFERENCES:
- [Background] Puechal X, Pagnoux C, Baron G, Quemeneur T, Neel A, Agard C, Lifermann F, Liozon E, Ruivard M, Godmer P, Limal N, Mekinian A, Papo T, Ruppert AM, Bourgarit A, Bienvenu B, Geffray L, Saraux JL, Diot E, Crestani B, Delbrel X, Sailler L, Cohen P, Le Guern V, Terrier B, Groh M, Le Jeunne C, Mouthon L, Ravaud P, Guillevin L; French Vasculitis Study Group. Adding Azathioprine to Remission-Induction Glucocorticoids for Eosinophilic Granulomatosis With Polyangiitis (Churg-Strauss), Microscopic Polyangiitis, or Polyarteritis Nodosa Without Poor Prognosis Factors: A Randomized, Controlled Trial. Arthritis Rheumatol. 2017 Nov;69(11):2175-2186. doi: 10.1002/art.40205. Epub 2017 Oct 15. PMID 28678392
- [Derived] Puechal X, Pagnoux C, Baron G, Lifermann F, Geffray L, Quemeneur T, Saraux JL, Wislez M, Cottin V, Ruivard M, Limal N, Aouba A, Bonnotte B, Neel A, Agard C, Cohen P, Terrier B, Le Jeunne C, Mouthon L, Ravaud P, Guillevin L; French Vasculitis Study Group investigators. Non-severe eosinophilic granulomatosis with polyangiitis: long-term outcomes after remission-induction trial. Rheumatology (Oxford). 2019 Dec 1;58(12):2107-2116. doi: 10.1093/rheumatology/kez139. PMID 31056661
- See also: Website of the French Vasculitis Study Group — http://www.vascularites.org